CLINICAL TRIAL: NCT03898466
Title: The Effect of Once-daily Fluticasone Furoate on Methacholine-induced Bronchoconstriction in Mild Asthmatics
Brief Title: Effect of Fluticasone Furoate on Methacholine Challenge
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Don Cockcroft, Professor, University of Saskatchewan
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Bio ID 366
Record Dates: First submitted 2019-03-29; First posted 2019-04-02 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — fluticasone furoate; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluticasone Furoate (Experimental): Daily inhalation of 100mcg fluticasone furoate for 7 days Response to methacholine induced bronchoconstriction will be assessed on Day 1 before first inhalation of study treatment (baseline) and again at 24, 72 and 168 hours.
  The change in airway responsiveness to methacholine will be determined as a dose shift in methacholine PD20 from baseline to each of the three timepoints
  Interventions: Drug: Fluticasone furoate
- Matching Placebo (Placebo Comparator): Daily inhalation of inactive placebo comparator for 7 days Response to methacholine induced bronchoconstriction will be assessed on Day 1 before first inhalation of study treatment (baseline) and again at 24, 72 and 168 hours.
  The change in airway responsiveness to methacholine will be determined as a dose shift in methacholine PD20 from baseline to each of the three timepoints
  Interventions: Other: Matching placebo

INTERVENTIONS:
Drug: Fluticasone furoate — Inhaled corticosteroid
  Other Names: Arnuity
  Arms: Fluticasone Furoate
Other: Matching placebo — Placebo inhaler
  Arms: Matching Placebo

SUMMARY:
The study will determine the effect of inhaled fluticasone furoate on airway responsiveness to methacholine in mild asthmatics.

ELIGIBILITY:
Inclusion Criteria:

* forced expiratory volume in one second (FEV1) greater than or equal to 65% predicted
* methacholine PD20 less than or equal to 400mcg
* no allergen exposure (if atopic) or respiratory infection for at least 4 weeks prior to study start

Exclusion Criteria:

* regular use of inhaled corticosteroid within 4 weeks of study start
* poorly controlled asthma
* current smoker or ex smoker with greater than 10 pack year history
* pregnancy or breast-feeding
* health concern/condition that would preclude participation for safety reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Methacholine provocation dose causing a 20% fall in FEV1 (PD20) | 24 hours post dose, 72 hours post dose and 168 hours post dose
  Change from baseline in airway response to inhaled methacholine following daily dosing with fluticasone furoate or placebo

SECONDARY OUTCOMES:
Fractional exhaled nitric oxide (FeNO) | 168 hours
  Change from baseline on levels of fractional exhaled nitric oxide
Sputum eosinophils | Baseline
  Assessment of induced sputum differential cell counts

CONTACTS AND LOCATIONS:
Locations (1):
- Asthma Research Lab University of Saskatchewan Room 346 Ellis Hall, Saskatoon, Saskatchewan, Canada

REFERENCES:
- [Derived] Okonkwo CS, Davis BE, Blais CM, Cockcroft DW. Short-term effect of once-daily fluticasone furoate on methacholine-induced bronchoconstriction in mild asthmatics. Respir Med. 2019 Sep;156:53-57. doi: 10.1016/j.rmed.2019.08.007. Epub 2019 Aug 13. PMID 31434037